CLINICAL TRIAL: NCT06254677
Title: Western Sydney Kidney Injury Biopsy Study
Acronym: WESTKiD
Status: Not yet recruiting | Type: Observational
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Jennifer Li, CPI, Nephrologist and Transplant Physician, Western Sydney Local Health District
Other Study IDs: WESTKiD
Record Dates: First submitted 2024-02-03; First posted 2024-02-12 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Access to histology slides: These slides are stored in the anatomical pathology department at Westmead Hospital/NSW Health Pathology. We will digitally scan these slides. Digital slides will be labelled with the study ID. Slides will be returned after scanning.
  Request access to kidney tissue blocks: This includes formalin-fixed, paraffin embedded (FFPE) kidney blocks, and fresh frozen kidney embedded in OCT. These are requested after clinical use and interpretation of the biopsy has been completed. The exact methodology will be determined by the available technology at the time (there is rapid advancement in imaging and molecular technologies) and the utility to achieve the objectives in the study. These include, but not limited to preparing slides for spatial transcriptomics (RNA-sequencing), single-cell extraction and RNA sequencing, spatial proteinomics, mass spectrometry/proteinomics, high plex immunohistochemistry, imaging mass cytometry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acute tubular injury (ATI) only: Kidney biopsy with features of acute tubular injury only, no other pathology detected
  Interventions: Other: Retrospective review of histological features
- Concurrent diagnosis of acute tubular injury with any other pathology: Kidney biopsy with features of acute tubular injury AND other pathology. Non-ATI pathology includes but not limited to diagnosis of any type of glomerulonephritis, vasculitis, hereditary nephritis, thrombotic microangiopathy, kidney transplant rejection, podocytopathy, diabetic or hypertensive nephropathy, interstitial nephritis, pyelonephritis, amyloidosis, malignancy or paraneoplastic related kidney disease.
  Interventions: Other: Retrospective review of histological features
- Biopsies with no acute tubular injury (neg control): Kidney biopsy with any diagnosis other than (no features of) acute tubular injury
  Interventions: Other: Retrospective review of histological features

INTERVENTIONS:
Other: Retrospective review of histological features — Correlate histopathology characteristics of acute kidney injury with molecular signatures, kidney function and aetiology of acute kidney injury to derive clinically validated scoring system for acute kidney injury and acute tubular injury

SUMMARY:
The investigators aim to develop a clinically validated, histological acute tubular injury (ATI) scoring system to help improve diagnostic precision and predict clinical outcomes following ATI.

To use an unbiased, data-driven approach, correlating pathological features (including digital pathology), key signatures using spatial technologies (transcriptomics or proteinomics) with relevant clinical outcomes. Spatial technologies (including spatial transcriptomics and spatial proteinomics) allow the use of 'precision pathology' to study the critical link between molecular characteristics to histological structure.

DETAILED DESCRIPTION:
The study is an investigator-led, retrospective, observational cohort study. This study is intended to be in perpetuity and there will be regular reporting to the local HREC (Western Sydney Local Health District, WSLHD)

Primary aim: the investigators aim to derive a clinically validated scoring system for acute kidney injury and iteratively improve its performance through machine learning algorithms over time.

Secondary aims:

* Derive a spatially resolved transcriptomic signature of acute kidney injury (AKI)
* Derive accurate transcriptomic signatures aligned with key cell types in AKI
* Derive unique gene signatures to differentiate different causes of AKI

All participants included in the study must be age ≥ 18 years old at time of enrolment and

1. Had a kidney transplant at any time after the year 2000
2. Kidney biopsy sample sent to Westmead Hospital for clinical interpretation
3. Have information regarding kidney function available.

This will include groups with

1. Acute tubular injury (ATI) only
2. ATI concurrently diagnosed with any other pathology on biopsy
3. Biopsies with no ATI (negative control)

Collection of health related data will be through review of primary medical records to improve the diagnostic utility of kidney biopsies performed to evaluate the cause of AKI.

The investigators will also be requesting waiver of consent for access to histopathology slides and residual kidney tissue

* Histopathology slides, which were created and analysed as part of routine clinical care.
* Residual kidney tissue, either as paraffin blocks or fresh frozen tissue

ELIGIBILITY:
Inclusion Criteria:

1. Had a kidney biopsy (native kidney or transplant kidney included) after year 2000
2. Kidney biopsy sample sent to Westmead Hospital for clinical interpretation

Exclusion Criteria:

1. Patients who have never had a kidney biopsy performed
2. Biopsy sample not available at Westmead Hospital
3. No information on kidney function (serum creatinine or eGFR)

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who had a kidney biopsy performed for any clinical indication, with biopsy sample sent to Westmead Hospital for review
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2035-01-01 (Estimated); Study Completion 2040-01-01 (Estimated)

PRIMARY OUTCOMES:
Histopathology characteristics of acute tubular injury (ATI) | Specific for the biopsy/tissue, no time frame after
  Biopsy features including tubular dilatation, interstitial oedema, epithelial vacuolization and disrupted brush border integrity
Kidney function | At biopsy (time 0) or during study follow up after biopsy (expected average 12-months)
  Kidney function based on blood tests collected from routine clinical care
Correlation of biopsy findings with kidney function at time of biopsy and longitudinally | At biopsy (time 0) or during study follow up after biopsy (expected average 12-months)
  Molecular signatures of injury

SECONDARY OUTCOMES:
Surrogate end point of kidney function | During study follow up after biopsy (expected average 12-months)
  eGFR slope
Albuminuria | At biopsy (time 0) or during study follow up after biopsy (expected average 12-months)
  urine albumin to creatinine ratio
Time to renal recovery | At biopsy (time 0) or during study follow up after biopsy (expected average 12-months)
  Kidney function return to baseline - based on any historical results before the biopsy date
Time to kidney failure | At biopsy (time 0) or during study follow up after biopsy (expected average 12-months)
  Deterioration (or no recovery) in kidney function where dialysis or transplantation is needed to sustain life
Chronic kidney disease | At biopsy (time 0) or during study follow up after biopsy (expected average 12-months)
  Deterioration (or without full recovery) in kidney function where chronic kidney disease is diagnosed based on clinical criteria
Response to treatment | At biopsy (time 0) or during study follow up after biopsy (expected average 12-months)
  Response to non-supportive therapy (eg steroids)
Genomic signatures | At biopsy (time 0) or during study follow up after biopsy (expected average 12-months)
  Transcriptomics (RNA) and microRNA (miRNA) extracted from the kidney biopsy
Cell types | At biopsy (time 0) or during study follow up after biopsy (expected average 12-months)
  Detection of immune or kidney cell types on kidney biopsy

IPD SHARING:
Plan to Share IPD: No